CLINICAL TRIAL: NCT06447922
Title: Analysis of Metal Ion Concentrations After Robotic-assisted Total Knee Arthroplasty Compared to Conventional Total Knee Arthroplasty
Brief Title: Metal Ion Concentrations After Total Knee Arthroplasty
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew P. Abdel, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 24-004661
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Arthroplasty, Replacement, Knee; Total Knee Replacement; Blood Metal Ion Concentration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Conventional TKA with Cutting Guides: Patients undergoing a conventional total knee arthroplasty with cutting guides (no robot-assistance).
  Interventions: Other: Metal ion level testing
- Robot-Assisted TKA: Patients undergoing a robot-assisted total knee arthroplasty.
  Interventions: Other: Metal ion level testing

INTERVENTIONS:
Other: Metal ion level testing — Patients will undergo a pre- and post-operative blood draw to analyze metal ion levels (Cobalt, Chromium, Titanium and Nickel)

SUMMARY:
The purpose of this study is to analyze the metal ion concentrations in the patients blood following robotic-assisted total knee arthroplasty (TKA) compared to conventional total knee arthroplasty using cutting guides.

DETAILED DESCRIPTION:
This study focuses on comparing metal ion levels in 50 inpatient participants undergoing primary total knee arthroplasty (TKA) with either conventional cutting guides or robotic assistance. Baseline blood examinations for Cobalt, Chromium, Titanium, and Nickel will be performed before TKA implantation at preoperative visits and on the first day following the procedure. The investigation will encompass patients receiving both conventional and robotic-assisted primary TKA, framed within a prospective cohort study design. Baseline characteristics and additional follow-up information will be gathered.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing conventional or robotic-assisted TKA
* Consent to the study

Exclusion Criteria:

* Patients who have undergone any previous arthroplasty procedures.
* Patients with metal implants, such as plates, nails, and screws, used in the repair of traumatic injuries.
* Patients below 110 pounds.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients eligible for a primary total knee replacement who have not had a prior joint replacement or surgery where metal implants were placed.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Overall blood metal ion differences between procedures (Conventional TKA vs Robot-Assisted TKA) | Pre-operatively, first post-operative day.
  Difference in overall blood metal ion levels (Cobalt, Chromium, Titanium, and Nickel) between patients undergoing total knee arthroplasty (TKA) with conventional cutting guides and those undergoing TKA with robotic assistance.

SECONDARY OUTCOMES:
Comparison of post-operative blood metal levels between procedures: Cobalt | First post-operative day
  Difference in post-operative levels, adjusted for the pre-operative levels, between Conventional TKA with Cutting Guides vs Robot-Assisted TKA
Comparison of post-operative blood metal levels between procedures: Chromium | First post-operative day
  Difference in post-operative levels, adjusted for the pre-operative levels, between Conventional TKA with Cutting Guides vs Robot-Assisted TKA
Comparison of post-operative blood metal levels between procedures: Titanium | First post-operative day
  Difference in post-operative levels, adjusted for the pre-operative levels, between Conventional TKA with Cutting Guides vs Robot-Assisted TKA
Comparison of post-operative blood metal levels between procedures: Nickel | First post-operative day
  Difference in post-operative levels, adjusted for the pre-operative levels, between Conventional TKA with Cutting Guides vs Robot-Assisted TKA

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Abdel, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No